CLINICAL TRIAL: NCT01496521
Title: Chemoprevention of Esophageal Squamous Cell Carcinoma With Aspirin and Tea Polyphenols: a Randomized Controlled Trial.
Brief Title: Chemoprevention of Esophageal Squamous Cell Carcinoma (ESCC) With Aspirin and Tea Polyphenols
Acronym: CREAT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Shu-Tian Zhang, Professor, Beijing Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CREAT
Record Dates: First submitted 2011-12-15; First posted 2011-12-21 (Estimated); Last update posted 2011-12-21 (Estimated); Status verified 2011-12

CONDITIONS: Carcinoma, Squamous Cell
Keywords: Aspirin; polyphenols; Chemoprevention
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Aspirin (Experimental)
  Interventions: Drug: Aspirin
- Tea Polyphenols (Experimental)
  Interventions: Dietary Supplement: Tea Polyphenols
- Control (No Intervention)

INTERVENTIONS:
Drug: Aspirin — 100mg qd for 6 months.
  Arms: Aspirin
Dietary Supplement: Tea Polyphenols — 300mg bid for 6 months.
  Arms: Tea Polyphenols

SUMMARY:
Evidence from laboratory studies suggests that aspirin and tea polyphenols may have an antineoplastic effect in esophageal squamous cell carcinoma (ESCC). To assess the safety and efficacy of aspirin and tea polyphenols for preventing ESCC, the investigators designed this double-blind, randomized controlled clinical trial. Research project is planned to recruit 10,000 participants with the ages of 40-60 years in Fengfeng city, Hebei province, China, which has been known as a high incidence region of ESCC. All the participants receive endoscopic examination. Lugol's chromoendoscopy is used to identify esophageal unstained lesions (USLs). The location and size of each USL will be recorded followed by collecting biopsy samples from each USL. Participants with USL are randomly assigned to receive 100 mg/d of aspirin (n=200), 100 mg/d of tea polyphenols (n=200), or placebo (n=200) for six months. Follow-up consists of 2 endoscopic surveillance cycles (the first interval will be at six months and the second at 3 or 5 years later). The primary outcome measure was occurrence of high grade dysplasia and invasive ESCC. Secondary outcome was the mortality of the participants and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. age 40 to 60 years;
2. Lugol's chromoendoscopy showing at least one USL 1 cm or larger containing mild to moderate dysplasia and chronic inflammation;
3. subject neither pregnant nor intending to become pregnant during the study.

Exclusion Criteria:

1. current non-steroidal anti-inflammatory drugs (NSAID) therapy;
2. major intercurrent illness;
3. pregnancy;
4. invasive carcinoma;
5. any condition that could be worsened by aspirin or tea polyphenols.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-06 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
occurrence of high grade dysplasia and invasive ESCC | at six months

SECONDARY OUTCOMES:
the mortality of the participants | The first interval will be at six months and the second at 3 or 5 years later.
Number of participants with adverse events. | The first interval will be at six months and the second at 3 or 5 years later.
occurrence of high grade dysplasia and invasive ESCC | at 3 or 5 years later

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Tian Zhang, MD, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital Capital Medical University, Beijing, China